CLINICAL TRIAL: NCT05045144
Title: A Phase III, Randomized, Multi-country Study to Evaluate the Lot-to-lot Consistency of GSK's Investigational RSV Maternal Vaccine and the Immune Response, Safety and Reactogenicity of RSV Maternal Vaccine When Co-administered With GSK's Quadrivalent Influenza D-QIV Vaccine in Healthy Non-pregnant Women 18-49 Years of Age.
Brief Title: A Phase III Study to Assess the Lot-to-lot Consistency of GSK's Investigational RSV Maternal Vaccine and the Immune Response and Safety of RSV Maternal Vaccine When Given Alone or Co-administered With GSK's Influenza D-QIV Vaccine in Healthy Non-pregnant Women.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 214709; 2021-000357-26 (EudraCT Number)
Record Dates: First submitted 2021-09-06; First posted 2021-09-16 (Actual); Results first posted 2023-10-05 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-09

CONDITIONS: Respiratory Syncytial Virus Infections
Keywords: Respiratory Syncytial Virus Maternal vaccine; Flu Quadrivalent influenza vaccine; Lot-to-lot consistency; Immunogenicity; Safety; Reactogenicity
MeSH Terms: conditions — Respiratory Syncytial Virus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Observer-blind (lot-to-lot consistency) & single-blind (immunogenicity, safety and reactogenicity)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- RSV lot1 Group (Experimental): Participants randomized to the RSV lot1 Group received one dose of RSV MAT Lot 1 vaccine intramuscularly at Day 1. Participants were also provided with an option of receiving Flu D-QIV vaccine at Day 31 to allow the participants receive the standard of care.
  Interventions: Combination Product: RSVPreF3(120 μg)
- RSV lot2 Group (Experimental): Participants randomized to the RSV lot2 Group received one dose of RSV MAT Lot 2 vaccine intramuscularly at Day 1. Participants were also provided with an option of receiving Flu D-QIV vaccine at Day 31 to allow the participants receive the standard of care.
  Interventions: Combination Product: RSVPreF3(120 μg)
- RSV lot3 Group (Experimental): Participants randomized to the RSV lot3 Group received one dose of RSV MAT Lot 3 vaccine intramuscularly at Day 1. Participants were also provided with an option of receiving Flu D-QIV vaccine at Day 31 to allow the participants receive the standard of care.
  Interventions: Combination Product: RSVPreF3(120 μg)
- RSV+Flu pooled Group (Experimental): Participants randomized in this group received one dose of RSVPreF3 vaccine (RSV MAT vaccine) from one of the three lots used (Lot 1, Lot 2 or Lot 3 of same formulation of RSVPreF3 vaccine) and one dose of the Flu D-QIV vaccine on Day 1, and were followed up until the end of the study (Day 181).
  The participants in this group were considered for the immunogenicity and safety analyses of the RSV MAT and Flu D-QIV vaccines.
  Interventions: Combination Product: Flu Quadrivalent influenza vaccine (15 μg HA)
- Flu+Placebo Group (Active Comparator): Participants randomized in this group received one dose of Flu D-QIV vaccine co-administered with one dose of placebo at Day 1, and were followed up until the end of the study (Day 181).
  This group was considered comparator for immunogenicity and safety analyses for RSV+ Flu Pooled group.
  Interventions: Combination Product: Flu Quadrivalent influenza vaccine (15 μg HA); Combination Product: Placebo

INTERVENTIONS:
Combination Product: RSVPreF3(120 μg) — A single dose of RSVPreF3(120 μg) combined with Sodium Chloride (NaCl) was administrated intramuscular (IM). There were used 3 different lots of RSVPreF3(120 μg), one for each individual group (RSV lot1 Group, RSV lot2 Group and RSV lot3 Group) considered under RSV pooled Group.
  Arms: RSV lot1 Group; RSV lot2 Group; RSV lot3 Group
Combination Product: Flu Quadrivalent influenza vaccine (15 μg HA) — A single dose of Flu Quadrivalent influenza (15 μg HA) vaccine was administrated intramuscular (IM).
  Arms: Flu+Placebo Group; RSV+Flu pooled Group
Combination Product: Placebo — One dose of placebo, administered intramuscularly in the deltoid region of the right arm, at Day 1.
  Arms: Flu+Placebo Group

SUMMARY:
The purpose of this study is to evaluate the clinical lot-to-lot consistency of the respiratory syncytial virus (RSV) maternal (RSV MAT) vaccine administered to healthy non-pregnant women 18-49 years of age (YOA). In addition, this study will evaluate immunogenicity, safety and reactogenicity from co-administration of RSV MAT vaccine and GSK's quadrivalent seasonal influenza (Flu D-QIV) vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Participants who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
* Written or witnessed/thumb printed informed consent obtained from the participant prior to performance of any study specific procedure.
* Healthy female participants; as established by medical history and clinical examination, aged 18 to 49 years at the time of the first study intervention administration.

  * Female participants of childbearing potential may be enrolled in the study, if the participant:
  * has practiced adequate contraception for 1 month prior to study intervention administration, and
  * has a negative pregnancy test on the day of study intervention administration, and
  * has agreed to continue adequate contraception during the entire treatment period and for 1 month after completion of the study intervention administration.
* No local condition precluding injection in both left and right deltoid muscles.

Exclusion Criteria:

Medical conditions

* History of any reaction or hypersensitivity likely to be exacerbated by any component of the study interventions;
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination;
* Current autoimmune disorder, for which the participant has received immune-modifying therapy within 6 months, before study vaccination;
* Hypersensitivity to latex;
* Acute or chronic clinically significant abnormality or poorly controlled pre-existent co-morbidities or any other clinical conditions, as determined by physical examination or medical history that, in the opinion of the investigator, might pose additional risk to the participant due to participation in the study;
* Significant or uncontrolled psychiatric illness;
* Recurrent history or uncontrolled neurological disorders or seizures;
* Documented HIV-positive participant;
* Body mass index > 40 kg/m^2;
* Any clinically significant* hematological parameter and/or biochemical laboratory abnormality.

  *The investigator should use his/her clinical judgment to decide which abnormalities are clinically significant.
* Any other clinical condition that, in the opinion of the investigator, might pose additional risk to the participant due to participation in the study.

Prior/Concomitant therapy

* Use of any investigational or non-registered product other than the study intervention(s) during the period starting 30 days before study intervention (Day -29 to Day 1), or planned use during the study period;
* Administration of long-acting immune-modifying drugs at any time during the study period;
* Administration of immunoglobulins and/or any blood products or plasma derivatives during the period starting 3 months before the study intervention or planned administration during the study period;
* Chronic administration of immunosuppressants or other immune-modifying drugs during the period starting 3 months prior to the first study intervention dose(s). For corticosteroids, this will mean prednisone 5 mg/day, or equivalent. Inhaled and topical steroids are allowed;
* Planned administration/administration of a vaccine not foreseen by the study protocol within the period starting 30 days before and ending 30 days after the vaccination dose;
* Administration of a seasonal influenza vaccine during the 6 months preceding entry into the study;
* Previous experimental vaccination against RSV.

Prior/Concurrent clinical study experience Concurrently participating in another clinical study, at any time during the study period, in which the participant has been or will be exposed to an investigational or a non-investigational vaccine/product;

Other exclusions

* Pregnant or lactating female;
* Female planning to become pregnant or planning to discontinue contraceptive precautions;
* Alcoholism or substance use disorder within the past 24 months based on the presence of two or more of the following abuse criteria: hazardous use, social/interpersonal problems related to use, neglected major roles to use, withdrawal tolerance, use of larger amounts or longer, repeated attempts to quit or control use, much time spent using, physical or psychological problems related to use, activities given up to use, craving;
* Any study personnel or their immediate dependents, family, or household members.

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Only healthy non-pregnant women 18-49 YOA are included in the study.
Enrollment: 1586 (Actual)
Dates: Start 2021-10-26 (Actual); Primary Completion 2022-06-06 (Actual); Study Completion 2022-06-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (31):
- United States (5):
  - GSK Investigational Site, West Palm Beach, Florida
  - GSK Investigational Site, Stockbridge, Georgia
  - GSK Investigational Site, Peoria, Illinois
  - GSK Investigational Site, Springfield, Missouri
  - GSK Investigational Site, Seattle, Washington
- Canada (11):
  - GSK Investigational Site, Surrey, British Columbia
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Truro, Nova Scotia
  - GSK Investigational Site, London, Ontario
  - GSK Investigational Site, Sarnia, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Mirabel, Quebec
  - GSK Investigational Site, Pointe-Claire, Quebec
  - GSK Investigational Site, Québec, Quebec
  - GSK Investigational Site, Saint-Charles-Borromée, Quebec
  - GSK Investigational Site, Sherbrooke, Quebec
- Finland (8):
  - GSK Investigational Site, Espoo
  - GSK Investigational Site, Helsinki
  - GSK Investigational Site, Jarvenpaa
  - GSK Investigational Site, Kokkola
  - GSK Investigational Site, Pori
  - GSK Investigational Site, Seinäjoki
  - GSK Investigational Site, Tampere
  - GSK Investigational Site, Turku
- South Korea (2):
  - GSK Investigational Site, Gyeonggi-do
  - GSK Investigational Site, Seoul
- Spain (5):
  - GSK Investigational Site, Alcorcón/Madrid
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Majadahonda (Madrid)
  - GSK Investigational Site, Santiago de Compostela
  - GSK Investigational Site, Valencia

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.

REFERENCES:
- [Derived] Chime N, Anspach B, Jain V, Laajalahti O, Ollinger T, Yaplee D, Kim JH. Phase 3 Study Assessing Lot-to-Lot Consistency of Respiratory Syncytial Virus Prefusion Protein F3 Vaccine and Its Immune Response, Safety, and Reactogenicity When Co-administered With Quadrivalent Influenza Vaccine. J Infect Dis. 2025 Feb 4;231(1):e144-e153. doi: 10.1093/infdis/jiae342. PMID 38970327

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Out of 1586 participants enrolled,47 participants did not receive vaccination as they did not meet the eligibility criteria or they were lost to follow up, therefore only 1539 participants were included in the Exposed Set and started the study.
Pre-assignment Details: As pre-specified in statistical plan, data reported in Participant Flow, Baseline Characteristics and Adverse Events were presented for individual RSV lot groups, pooled RSV+Flu group (since minimal differences were expected between participants who received different RSV lots of the vaccine) and Flu+Placebo Group. As pre-specified in protocol, immunogenicity outcome measures presented data for the pooled RSV and RSV+Flu groups, and individual RSV lot groups were used for lot-to-lot analyses.
Period: Overall Study
Arm/Group | RSV lot1 Group | RSV lot2 Group | RSV lot3 Group | RSV+Flu Pooled Group | Flu+Placebo Group
Started | 220 | 223 | 218 | 438 | 440
Completed | 217 | 220 | 214 | 433 | 427
Not Completed | 3 | 3 | 4 | 5 | 13
Not completed — Lost to Follow-up | 3 | 2 | 3 | 5 | 13
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0
Not completed — MIGRATED / MOVED FROM THE STUDY AREA | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RSV lot1 Group | RSV lot2 Group | RSV lot3 Group | RSV+Flu Pooled Group | Flu+Placebo Group | Total
Number analyzed (Participants) | 220 | 223 | 218 | 438 | 440 | 1539
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 32.0 (9.6) | 31.4 (9.4) | 31.9 (9.3) | 32.0 (8.9) | 32.1 (8.9) | 31.9 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 220 | 223 | 218 | 438 | 440 | 1539
  Male | 0 | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  AMERICAN INDIAN OR ALASKA NATIVE | 2 | 4 | 3 | 10 | 7 | 26
  ASIAN | 22 | 25 | 21 | 38 | 43 | 149
  BLACK OR AFRICAN AMERICAN | 12 | 3 | 6 | 17 | 17 | 55
  NATIVE HAWAIIAN OR OTHER PACIFIC ISLANDER | 0 | 0 | 0 | 1 | 0 | 1
  OTHER | 1 | 4 | 3 | 3 | 7 | 18
  WHITE | 183 | 187 | 185 | 369 | 366 | 1290

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Reporting Solicited Administration Site Events in RSV Pooled Group, RSV+Flu Pooled Group and Flu+Placebo Group
Description: Assessed solicited administration site events include pain, erythema and swelling. This objective analyzed the safety and reactogenicity of RSV MAT vaccine when given alone (pooled lots) or co-administered with Flu D-QIV. As pre-specified in protocol, data reported in this outcome measure was presented for the pooled RSV and RSV+Flu groups and Flu+Placebo Group, since minimal differences were expected between participants who received different RSV lots of the vaccine.
Time Frame: From Day 1 to Day 7 (including Day 7)
Population: Analysis was performed on the Solicited Safety Set (SSS), which includes all participants who received at least 1 dose of the study intervention (Exposed Set [ES]) and who have solicited safety data.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- RSV Pooled Group: Participants randomized in this group received one dose of RSVPreF3 vaccine (RSV MAT vaccine) on Day 1, from one of the three lots used (Lot 1, Lot 2 or Lot 3 of same formulation of RSVPreF3 vaccine) and were followed up until the end of the study (Day 181). On Day 31 (Visit 2), participants in this group had the option to receive the Flu D-QIV vaccine, as part of their standard of care.
  This group was considered for the immunogenicity and safety analysis of the RSV MAT vaccine.
Arm/Group | RSV Pooled Group | RSV+Flu Pooled Group | Flu+Placebo Group
Number analyzed (Participants) | 660 | 438 | 439
Percentage of participants
  Pain | 53.6 [49.7 to 57.5] | 51.1 [46.4 to 55.9] | 34.4 [30 to 39]
  Erythema | 4.4 [3 to 6.2] | 3.7 [2.1 to 5.9] | 0.5 [0.1 to 1.6]
  Swelling | 4.5 [3.1 to 6.4] | 4.6 [2.8 to 7] | 0.9 [0.2 to 2.3]

2. Primary Outcome: Percentage of Participants Reporting Solicited Systemic Events in RSV Pooled Group, RSV+Flu Pooled Group and Flu+Placebo Group
Description: Assessed solicited systemic events include fatigue, headache, gastrointestinal (GI) symptoms (nausea, vomiting, diarrhea, abdominal pain) and fever. The preferred location for measuring temperature was the oral cavity. Fever was defined as temperature equal to or above (≥) 38.0 °C/ 100.4°F. This objective analyzed the safety and reactogenicity of RSV MAT vaccine when given alone (pooled lots) or co-administered with Flu D-QIV. As pre-specified in protocol, data reported in this outcome measure was presented for the pooled RSV and RSV+Flu groups and Flu+Placebo Group, since minimal differences were expected between participants who received different RSV lots of the vaccine.
Time Frame: From Day 1 to Day 7 (including Day 7)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Groups:
- RSV Pooled Group: Participants randomized in this group received one dose of RSVPreF3 vaccine (RSV MAT vaccine) on Day 1, from one of the three lots used (Lot 1, Lot 2 or Lot 3 of same formulation of RSVPreF3 vaccine) and were followed up until the end of the study (Day 181). On Day 31 (Visit 2), participants in this group had the option to receive the Flu D-QIV vaccine per strain/dose, as part of their standard of care.
Arm/Group | RSV Pooled Group | RSV+Flu Pooled Group | Flu+Placebo Group
Number analyzed (Participants) | 660 | 438 | 439
Percentage of participants
  Fatigue | 52 [48.1 to 55.8] | 59.8 [55.1 to 64.4] | 51.9 [47.1 to 56.7]
  Headache | 47.6 [43.7 to 51.5] | 51.4 [46.6 to 56.1] | 43.1 [38.4 to 47.8]
  Nausea | 14.5 [11.9 to 17.5] | 15.3 [12.1 to 19] | 12.3 [9.4 to 15.7]
  Vomiting | 2.3 [1.3 to 3.7] | 1.8 [0.8 to 3.6] | 2.3 [1.1 to 4.1]
  Diarrhea | 12.1 [9.7 to 14.9] | 13 [10 to 16.5] | 17.1 [13.7 to 20.9]
  Abdominal pain | 12 [9.6 to 14.7] | 13.5 [10.4 to 17] | 14.1 [11 to 17.7]
  Temperature | 2.4 [1.4 to 3.9] | 3 [1.6 to 5] | 0.7 [0.1 to 2]

3. Primary Outcome: Percentage of Participants Reporting Unsolicited Adverse Events (AEs) in RSV Pooled Group, RSV+Flu Pooled Group and Flu+Placebo Group
Description: An unsolicited AE is any AE reported in addition to those solicited during the clinical study. Also, any 'solicited' symptom with onset outside the specified period of follow-up for solicited symptoms is reported as an unsolicited adverse event. This objective analyzed the safety and reactogenicity of RSV MAT vaccine when given alone (pooled lots) or co-administered with Flu D-QIV. As pre-specified in protocol, data reported in this outcome measure was presented for the pooled RSV and RSV+Flu groups and Flu+Placebo Group, since minimal differences were expected between participants who received different RSV lots of the vaccine.
Time Frame: From Day 1 to Day 30 (including Day 30)
Population: Analysis was performed on the ES (Exposed Set), which includes all participants who received at least 1 dose of the study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | RSV Pooled Group | RSV+Flu Pooled Group | Flu+Placebo Group
Number analyzed (Participants) | 661 | 438 | 440
Percentage of participants | 26.6 [23.3 to 30.2] | 30.1 [25.9 to 34.7] | 25.7 [21.7 to 30]

4. Primary Outcome: Percentage of Participants Reporting Serious Adverse Events (SAEs) in RSV Pooled Group, RSV+Flu Pooled Group and Flu+Placebo Group
Description: An SAE is any untoward medical occurrence that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study participant or results i+F2n abnormal pregnancy outcomes. This objective analyzed the safety and reactogenicity of RSV MAT vaccine when given alone (pooled lots) or co-administered with Flu D-QIV. As pre-specified in protocol, data reported in this outcome measure was presented for the pooled RSV and RSV+Flu groups and Flu+Placebo Group, since minimal differences were expected between participants who received different RSV lots of the vaccine.
Time Frame: From Day 1 to Day 30 (including Day 30)
Population: Analysis was performed on the ES, which includes all participants who received at least 1 dose of the study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | RSV Pooled Group | RSV+Flu Pooled Group | Flu+Placebo Group
Number analyzed (Participants) | 661 | 438 | 440
Percentage of participants | 0.2 [0 to 0.8] | 0 [0 to 0.8] | 0.2 [0 to 1.3]

5. Primary Outcome: Percentage of Participants Reporting SAEs in RSV Pooled Group, RSV+Flu Pooled Group and Flu+Placebo Group
Description: An SAE is any untoward medical occurrence that results in death, is life-threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect in the offspring of a study participant or results in abnormal pregnancy outcomes.This objective analyzed the safety and reactogenicity of RSV MAT vaccine when given alone (pooled lots) or co-administered with Flu D-QIV. As pre-specified in protocol, data reported in this outcome measure was presented for the pooled RSV and RSV+Flu groups and Flu+Placebo Group, since minimal differences were expected between participants who received different RSV lots of the vaccine.
Time Frame: From first vaccination up to study end (Day 1 to Day 181)
Population: Analysis is performed on the ES, which includes all participants who received at least 1 dose of the study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | RSV Pooled Group | RSV+Flu Pooled Group | Flu+Placebo Group
Number analyzed (Participants) | 661 | 438 | 440
Percentage of participants | 0.8 [0.2 to 1.8] | 0.9 [0.2 to 2.3] | 0.9 [0.2 to 2.3]

6. Primary Outcome: RSV MAT Immunoglobulin G (IgG) Enzyme-Linked Immunosorbent Assay (ELISA) Concentrations for Participants in RSV lot1, RSV lot2 and RSV lot3 Groups at Day 31
Description: Serological assays for the determination of IgG antibodies against RSV MAT were performed by ELISA. RSV MAT IgG concentrations were expressed as geometric mean concentrations (GMCs), in ELISA units per milliliter (EU/mL). As pre-specified in protocol, data reported in this outcome measure was presented only for individual RSV lot groups (RSV lot1, RSV lot2, RSV lot3), as the purpose was to analyze RSV MAT IgG ELISA concentrations, in order to demonstrate the lot-to-lot consistency of the vaccine lots.
Time Frame: At Day 31
Population: Analysis was performed on the Per Protocol Set (PPS), only on the participants who received only 1 dose of RSV MAT vaccine (from RSV MAT vaccine Lot 1, Lot 2 or Lot 3), and have post-vaccination data, from which are excluded participants with protocol deviations and for whom immunogenicity results were available for the specified assay and time point.
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | RSV lot1 Group | RSV lot2 Group | RSV lot3 Group
Number analyzed (Participants) | 201 | 204 | 207
EU/mL | 102811.0 [95243.6 to 110979.6] | 100635.8 [92970.2 to 108933.4] | 108709.3 [101913.7 to 115958.0]
Statistical Analysis 1: Comparison: RSV lot1 Group vs RSV lot2 Group; To demonstrate lot-to-lot consistency of the immune responses of Lot 1 and Lot 2 of the RSV MAT vaccine, as measured by ELISA in terms of IgG GMCs at Day 31; Test type: Other — The lot-to-lot consistency is demonstrated only if two-sided 95% confidence intervals (CI) for the 3 pair-wise geometric mean ratios of RSV MAT IgG ELISA concentration falls within 0.67 and 1.5; GMC ratio; GMC Ratio = 1.02, 95% CI 2-sided [0.92 to 1.13]
Statistical Analysis 2: Comparison: RSV lot1 Group vs RSV lot3 Group; To demonstrate lot-to-lot consistency of the immune responses of Lot 1 and Lot 3 of the RSV MAT vaccine, as measured by ELISA in terms of IgG GMCs at Day 31; Test type: Other — [test comment as in outcome 6, analysis 1]; GMC ratio; GMC ratio = 0.95, 95% CI 2-sided [0.85 to 1.05]
Statistical Analysis 3: Comparison: RSV lot2 Group vs RSV lot3 Group; To demonstrate lot-to-lot consistency of the immune responses of Lot 2 and Lot 3 of the RSV MAT vaccine, as measured by ELISA in terms of IgG GMCs at Day 31; Test type: Other — [test comment as in outcome 6, analysis 1]; GMC ratio; GMC ratio = 0.93, 95% CI 2-sided [0.83 to 1.03]

7. Primary Outcome: Flu D-QIV Haemagglutinin Inhibition (HI) Antibody Titers Against 3 Influenza Strains for Participants in Flu+Placebo Group and RSV+Flu Pooled Group at Day 31
Description: Flu D-QIV HI antibody titers against 3 influenza strains (A/Tasmania/503/2020 (H3N2) IVR-221; B/Washington/02/2019; B/Phuket/3073/2013) were expressed as geometric mean titers (GMTs), as assessed by HI assay. This objective analyzed the humoral immune response to the Flu D-QIV vaccine when given alone and co-administered with RSV MAT vaccine in terms of antibody titers against 3 influenza strains. As pre-specified in protocol, data reported in this outcome measure was presented for the pooled RSV+Flu Group and Flu+Placebo Group, since minimal differences were expected between participants who received different RSV lots of the vaccine.
Time Frame: At Day 31
Population: Analysis was performed on the Per Protocol Set (PPS), only on the participants who received 1 dose of Flu D-QIV vaccine and optionally other study treatment, and have post-vaccination data, from which are excluded participants with protocol deviations and for whom immunogenicity results were available for the specified assay and time point.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | RSV+Flu Pooled Group | Flu+Placebo Group
Number analyzed (Participants) | 398 | 404
Titers
  A/Tasmania/503/2020 (H3N2) | 301.6 [274.0 to 331.9] | 421.3 [383.4 to 463.0]
  B/Washington/02/2019 | 30.7 [27.3 to 34.6] | 33.0 [29.3 to 37.2]
  B/Phuket/3073/2013 | 56.2 [50.7 to 62.3] | 69.9 [62.6 to 77.9]
Statistical Analysis 1: Comparison: RSV+Flu Pooled Group vs Flu+Placebo Group; To demonstrate the immunological non-inferiority of the Flu D-QIV vaccine when co-administered with RSV MAT vaccine compared to Flu D-QIV vaccine given alone as measured by the ratio of HI GMTs of Flu D-QIV antibody titers against A/Tasmania/503/2020 (H3N2) IVR-221 strain at 30 days post administration (Day 31); Test type: Non-Inferiority — The non-inferiority of Flu D-QIV vaccine is demonstrated for the A/Tasmania/503/2020 (H3N2) IVR-221 strain, if the lower limit (LL) of the 95% CI on the GMT ratio (RSV MAT + Flu D-QIV vaccine divided by Flu D-QIV vaccine) is greater than 0.67 at Day 31 post vaccination; GMC ratio; GMC ratio = 0.72, 95% CI 2-sided [0.63 to 0.82]
Statistical Analysis 2: Comparison: RSV+Flu Pooled Group vs Flu+Placebo Group; To demonstrate the immunological non-inferiority of the Flu D-QIV vaccine when co-administered with RSV MAT vaccine compared to Flu D-QIV vaccine given alone as measured by the ratio of HI GMTs of Flu D-QIV antibody titers against B/Washington/02/2019 strain at 30 days post administration (Day 31); Test type: Non-Inferiority — The non-inferiority of Flu D-QIV vaccine is demonstrated for B/Washington/02/2019 strain, if the lower limit (LL) of the 95% CI on the GMT ratio (RSV MAT + Flu D-QIV vaccine divided by Flu D-QIV vaccine) is greater than 0.67 at Day 31 post vaccination; GMC ratio; GMC ratio = 0.93, 95% CI 2-sided [0.79 to 1.10]
Statistical Analysis 3: Comparison: RSV+Flu Pooled Group vs Flu+Placebo Group; To demonstrate the immunological non-inferiority of the Flu D-QIV vaccine when co-administered with RSV MAT vaccine compared to Flu D-QIV vaccine given alone as measured by the ratio of HI GMTs of Flu D-QIV antibody titers against B/Phuket/3073/2013 strain at 30 days post administration (Day 31); Test type: Non-Inferiority — The non-inferiority of Flu D-QIV vaccine is demonstrated for B/Phuket/3073/2013 strain, if the lower limit (LL) of the 95% CI on the GMT ratio (RSV MAT + Flu D-QIV vaccine divided by Flu D-QIV vaccine) is greater than 0.67 at Day 31 post vaccination; GMC ratio; GMC ratio = 0.80, 95% CI 2-sided [0.69 to 0.93]

8. Secondary Outcome: RSV A Neutralizing Antibody Titers for Participants in RSV Pooled Group and RSV+Flu Pooled Group at Day 1 and Day 31
Description: Serological assays for the determilnation of antibodies against RSV A were performed by neutralization assay. RSV A neutralizing antibody titers were expressed as geometric mean titers (GMTs), in serum dilution inducing 60% inhibition in plaque forming units (ED60). This objective analyzed the humoral immune response of RSV MAT vaccine when given alone and co-administered with Flu D-QIV in terms of RSV A neutralizing antibody. As pre-specified in protocol, data reported in this outcome measure was presented for the pooled RSV and RSV+Flu groups, since minimal differences were expected between participants who received different RSV lots of the vaccine.
Time Frame: At Day 1 and Day 31
Population: Analysis was performed on the Per Protocol Set (PPS), only on the participants who received 1 dose of RSV MAT vaccine (from one of the 3 lots used) and optionally other study treatment, and have post-vaccination data, from which are excluded participants with protocol deviations and for whom immunogenicity results were available for the specified assay and time point.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | RSV Pooled Group | RSV+Flu Pooled Group
Number analyzed (Participants) | 657 | 436
Titers
  Day 1 | 721.6 [676.5 to 769.7] | 707.2 [653.4 to 765.5]
  Day 31: number analyzed (Participants) | 611 | 398
  Day 31 | 8900.9 [8272.1 to 9577.5] | 7761.6 [7092.8 to 8493.6]
Statistical Analysis 1: Comparison: RSV Pooled Group vs RSV+Flu Pooled Group; To demonstrate the immunological non-inferiority of the RSV MAT vaccine when co-administered with Flu D-QIV vaccine, compared to RSV MAT vaccine given alone as measured by the ratio of GMTs of RSV A neutralizing antibody titers at 30 days post administration (Day 31); Test type: Non-Inferiority — The non-inferiority of RSV MAT vaccine is demonstrated for RSV A neutralizing antibody titers, if the LL of the 95% CI on the GMT ratio (RSV MAT + Flu D-QIV vaccine divided by RSV MAT vaccine) is greater than 0.67 at Day 31 post vaccination; GMC ratio; GMC ratio = 0.87, 95% CI 2-sided [0.78 to 0.97]

9. Secondary Outcome: Seroconversion Rate (SCR) to Flu D-QIV HI Antibody Titers Against 3 Influenza Strains for Participants in Flu+Placebo Group and RSV+Flu Pooled Group at Day 31
Description: The SCR was defined as the percentage of participants with: a Day 1 (pre-vaccination) serum anti-HI titer <1:10 and a Day 31 (post-vaccination) serum anti-HI titer ≥1:40, or a Day 1 (pre-vaccination) serum anti-HI titer ≥ 1:10 and a fold increase (post/pre) ≥ 4 at Day 31. The 3 influenza strains assessed were: A/Tasmania/503/2020 (H3N2) IVR-221; B/Washington/02/2019 and B/Phuket/3073/2013. This objective analyzed the seroconversion rate to the Flu D-QIV vaccine when given alone and co-administered with RSV MAT vaccine. As pre-specified in protocol, data reported in this outcome measure was presented for the pooled RSV+Flu group and Flu+Placebo Group, since minimal differences were expected between participants who received different RSV lots of the vaccine.
Time Frame: At Day 31
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | RSV+Flu Pooled Group | Flu+Placebo Group
Number analyzed (Participants) | 398 | 403
Percentage of participants
  A/Tasmania/503/2020 (H3N2) | 42.5 [37.6 to 47.5] | 45.9 [41 to 50.9]
  B/Washington/02/2019 | 25.4 [21.2 to 30] | 29.5 [25.1 to 34.2]
  B/Phuket/3073/2013 | 31.4 [26.9 to 36.2] | 35.5 [30.8 to 40.4]
Statistical Analysis 1: Comparison: RSV+Flu Pooled Group vs Flu+Placebo Group; To demonstrate the immunological non-inferiority of the Flu D-QIV vaccine when co-administered with RSV MAT vaccine compared to Flu D-QIV vaccine given alone as measured by the difference of proportion of participants achieving seroconversion for HI antibody titers against A/Tasmania/503/2020 (H3N2) IVR-221 strain at 30 days post administration (Day 31); Test type: Non-Inferiority — The non-inferiority of Flu D-QIV vaccine is demonstrated with respect to the SCR difference for Flu D-QIV antibody titers against A/Tasmania/503/2020 (H3N2) IVR-221 strain, if the upper limit (UL) of the 95% CI on the SCR difference (Flu D-QIV vaccine minus RSV MAT + Flu D-QIV vaccine) is less than or equal to the pre-defined clinical limit of 10% at Day 31 post vaccination; Miettinen and Nurminen; Difference of Proportion = 3.44, 95% CI 2-sided [-3.44 to 10.29]
Statistical Analysis 2: Comparison: RSV+Flu Pooled Group vs Flu+Placebo Group; To demonstrate the immunological non-inferiority of the Flu D-QIV vaccine when co-administered with RSV MAT vaccine compared to Flu D-QIV vaccine given alone as measured by the difference of proportion of participants achieving seroconversion for HI antibody titers against B/Washington/02/2019 strain at 30 days post administration (Day 31); Test type: Non-Inferiority — The non-inferiority of Flu D-QIV vaccine is demonstrated with respect to the SCR difference for Flu D-QIV antibody titers against B/Washington/02/2019 strain, if the upper limit (UL) of the 95% CI on the SCR difference (Flu D-QIV vaccine minus RSV MAT + Flu D-QIV vaccine) is less than or equal to the pre-defined clinical limit of 10% at Day 31 post vaccination; Miettinen and Nurminen; Difference of Proportion = 4.15, 95% CI 2-sided [-2.04 to 10.32]
Statistical Analysis 3: Comparison: RSV+Flu Pooled Group vs Flu+Placebo Group; To demonstrate the immunological non-inferiority of the Flu D-QIV vaccine when co-administered with RSV MAT vaccine compared to Flu D-QIV vaccine given alone as measured by the difference of proportion of participants achieving seroconversion for HI antibody titers against B/Phuket/3073/2013 strain at 30 days post administration (Day 31); Test type: Non-Inferiority — The non-inferiority of Flu D-QIV vaccine is demonstrated with respect to the SCR difference for Flu D-QIV antibody titers against B/Phuket/3073/2013 strain, if the upper limit (UL) of the 95% CI on the SCR difference (Flu D-QIV vaccine minus RSV MAT + Flu D-QIV vaccine) is less than or equal to the pre-defined clinical limit of 10% at Day 31 post vaccination; Miettinen and Nurminen; Difference of Proportion = 4.08, 95% CI 2-sided [-2.46 to 10.58]

10. Secondary Outcome: RSV B Neutralizing Antibody Titers for Participants in RSV Pooled Group and RSV+Flu Pooled Group at Day 1 and Day 31
Description: Serological assays for the determination of antibodies against RSV B were performed by neutralization assay. RSV B neutralizing antibody titers were expressed as GMTs, in ED60. This objective analyzed the humoral immune response of RSV MAT vaccine when given alone and co-administered with Flu D-QIV in terms of RSV B neutralizing antibody. As pre-specified in protocol, data reported in this outcome measure was presented for the pooled RSV and RSV+Flu groups, since minimal differences were expected between participants who received different RSV lots of the vaccine.
Time Frame: At Day 1 and Day 31
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | RSV Pooled Group | RSV+Flu Pooled Group
Number analyzed (Participants) | 656 | 436
Titers
  Day 1 | 967.4 [909.5 to 1028.9] | 940.1 [871 to 1014.6]
  Day 31: number analyzed (Participants) | 610 | 398
  Day 31 | 11030.5 [10344.5 to 11762] | 9162.3 [8483.3 to 9895.8]

11. Secondary Outcome: RSV MAT IgG Concentrations for Participants in RSV Pooled Group and RSV+Flu Pooled Group at Day 1 and Day 31
Description: Serological assays for the determination of IgG antibodies against RSV MAT were performed by ELISA. RSV MAT IgG concentrations were expressed as GMCs, in EU/mL. This objective analyzed the humoral immune response of RSV MAT vaccine when given alone and co-administered with Flu D-QIV in terms of RSV MAT IgG concentrations. As pre-specified in protocol, data reported in this outcome measure was presented for the pooled RSV and RSV+Flu groups, since minimal differences were expected between participants who received different RSV lots of the vaccine.
Time Frame: At Day 1 and Day 31
Population: as for outcome 8
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | RSV Pooled Group | RSV+Flu Pooled Group
Number analyzed (Participants) | 657 | 436
EU/mL
  Day 1 | 5522.7 [5285.7 to 5770.4] | 5772 [5455.8 to 6106.4]
  Day 31: number analyzed (Participants) | 612 | 398
  Day 31 | 104025.1 [99714.5 to 108522.2] | 83937 [79640.9 to 88464.9]

12. Secondary Outcome: Flu D-QIV HI Antibody Titers Against 3 Influenza Strains for Participants in Flu+Placebo Group and RSV+Flu Pooled Group at Day 1 and Day 31
Description: Flu D-QIV HI antibody titers against 3 influenza strains (A/Tasmania/503/2020 (H3N2) IVR-221;B/Washington/02/2019; B/Phuket/3073/2013) were expressed as geometric mean titers (GMTs), as assessed by HI assay. This objective analyzed the humoral immune response to the Flu D-QIV vaccine when given alone and co-administered with RSV MAT vaccine in terms of antibody titers against 3 influenza strains. As pre-specified in protocol, data reported in this outcome measure was presented for the pooled RSV+Flu Group and Flu+Placebo Group, since minimal differences were expected between participants who received different RSV lots of the vaccine.
Time Frame: At Day 1 and Day 31
Population: as for outcome 7
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | RSV+Flu Pooled Group | Flu+Placebo Group
Number analyzed (Participants) | 436 | 437
Titers
  A/Tasmania/503/2020 (H3N2) , Day 1 | 92.2 [81.2 to 104.8] | 110.3 [97.2 to 125.1]
  A/Tasmania/503/2020 (H3N2) , Day 31: number analyzed (Participants) | 398 | 404
  A/Tasmania/503/2020 (H3N2) , Day 31 | 301.6 [274 to 331.9] | 421.3 [383.4 to 463]
  B/Washington/02/2019 , Day 1 | 11.7 [10.6 to 13] | 10.3 [9.4 to 11.3]
  B/Washington/02/2019 , Day 31: number analyzed (Participants) | 398 | 404
  B/Washington/02/2019 , Day 31 | 30.7 [27.3 to 34.6] | 33 [29.3 to 37.2]
  B/Phuket/3073/2013 , Day 1 | 21.2 [19 to 23.7] | 21.9 [19.6 to 24.5]
  B/Phuket/3073/2013 , Day 31: number analyzed (Participants) | 398 | 404
  B/Phuket/3073/2013 , Day 31 | 56.2 [50.7 to 62.3] | 69.9 [62.6 to 77.9]

13. Secondary Outcome: Seroprotection Rate (SPR) to Flu D-QIV HI Antibody Titers for Participants in Flu+Placebo Group and RSV+Flu Pooled Group at Day 1 and Day 31
Description: SPR was measured by the percentage of participants achieving an HI antibody titer ≥1:40. This objective analyzed the seroprotection rate to the Flu D-QIV vaccine when given alone and co-administered with RSV MAT vaccine. As pre-specified in protocol, data reported in this outcome measure was presented for the pooled RSV+Flu Group and Flu+Placebo Group, since minimal differences were expected between participants who received different RSV lots of the vaccine.
Time Frame: At Day 1 and Day 31
Population: as for outcome 7
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | RSV+Flu Pooled Group | Flu+Placebo Group
Number analyzed (Participants) | 436 | 437
Percentage of participants
  A/Tasmania/503/2020 (H3N2) , Day 1 | 78.7 [74.5 to 82.4] | 82.8 [79 to 86.3]
  A/Tasmania/503/2020 (H3N2) , Day 31: number analyzed (Participants) | 398 | 404
  A/Tasmania/503/2020 (H3N2) , Day 31 | 98 [96.1 to 99.1] | 98.5 [96.8 to 99.5]
  B/Washington/02/2019 , Day 1 | 19.7 [16.1 to 23.8] | 16.9 [13.5 to 20.8]
  B/Washington/02/2019 , Day 31: number analyzed (Participants) | 398 | 404
  B/Washington/02/2019 , Day 31 | 48 [43 to 53] | 48.8 [43.8 to 53.8]
  B/Phuket/3073/2013 , Day 1 | 36.7 [32.2 to 41.4] | 39.8 [35.2 to 44.6]
  B/Phuket/3073/2013 , Day 31: number analyzed (Participants) | 398 | 404
  B/Phuket/3073/2013 , Day 31 | 74.4 [69.8 to 78.6] | 77.2 [72.8 to 81.2]

14. Secondary Outcome: RSV A Neutralizing Antibody Titers for Participants in RSV lot1, RSV lot2 and RSV lot3 Groups at Day 1 and Day 31
Description: Serological assays for the determination of antibodies against RSV-A were performed by neutralization assay. RSV A neutralizing antibody titers were expressed as GMTs, in ED60. As pre-specified in protocol, data reported in this outcome measure was presented only for individual RSV lot groups (RSV lot1, RSV lot2, RSV lot3), as the purpose was to analyze the humoral immune response of RSV A neutralizing antibody titers, in order to demonstrate the lot-to-lot consistency of the vaccine lots.
Time Frame: At Day 1 and Day 31
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | RSV lot1 Group | RSV lot2 Group | RSV lot3 Group
Number analyzed (Participants) | 217 | 223 | 217
Titers
  Day 1 | 727.5 [652 to 811.6] | 758.4 [676.7 to 849.9] | 680.2 [607.4 to 761.7]
  Day 31: number analyzed (Participants) | 201 | 204 | 206
  Day 31 | 8545.5 [7464.4 to 9783.2] | 8760.3 [7716.2 to 9945.8] | 9409.2 [8343.5 to 10611]

15. Secondary Outcome: RSV B Neutralizing Antibody Titers for Participants in RSV lot1, RSV lot2 and RSV lot3 Groups at Day 1 and Day 31
Description: Serological assays for the determination of antibodies against RSV B were performed by neutralization assay. RSV B neutralizing antibody titers were expressed as GMTs, in ED60. As pre-specified in protocol, data reported in this outcome measure was presented only for individual RSV lot groups (RSV lot1, RSV lot2, RSV lot3), as the purpose was to analyze the humoral immune response of RSV B neutralizing antibody titers, in order to demonstrate the lot-to-lot consistency of the vaccine lots.
Time Frame: At Day 1 and Day 31
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | RSV lot1 Group | RSV lot2 Group | RSV lot3 Group
Number analyzed (Participants) | 216 | 223 | 217
Titers
  Day 1 | 895 [810.6 to 988.2] | 1030.3 [929.3 to 1142.3] | 979.7 [870.6 to 1102.4]
  Day 31: number analyzed (Participants) | 201 | 204 | 205
  Day 31 | 10457 [9258.5 to 11810.6] | 11107.2 [9984.4 to 12356.4] | 11543.3 [10377.6 to 12840.1]

16. Secondary Outcome: RSV MAT IgG Concentrations for Participants in RSV lot1, RSV lot2 and RSV lot3 Groups at Day 1 and Day 31
Description: Serological assays for the determination of IgG antibodies against RSV MAT were performed by ELISA. RSV MAT IgG concentrations were expressed as GMCs, in EU/mL. As pre-specified in protocol, data reported in this outcome measure was presented only for individual RSV lot groups (RSV lot1, RSV lot2, RSV lot3), as the purpose was to analyze the RSV MAT IgG concentration, in order to demonstrate the lot-to-lot consistency of the vaccine lots.
Time Frame: At Day 1 and Day 31
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | RSV lot1 Group | RSV lot2 Group | RSV lot3 Group
Number analyzed (Participants) | 217 | 223 | 217
EU/mL
  Day 1 | 5691.9 [5276.8 to 6139.7] | 5613 [5197.8 to 6061.3] | 5270.1 [4883.6 to 5687.1]
  Day 31: number analyzed (Participants) | 201 | 204 | 207
  Day 31 | 102811 [95243.6 to 110979.6] | 100635.8 [92970.2 to 108933.4] | 108709.3 [101913.7 to 115958]

ADVERSE EVENTS:
Time Frame: Serious Adverse Events (SAEs) were collected through the entire period of the study (from Day 1 up to study end [Day 181]). Solicited AEs were collected from Day 1 to Day 7 included and unsolicited AEs were collected from Day 1 to Day 30 included.
Description: As pre-specified in protocol, adverse events were presented for individual RSV lot groups, RSV+Flu pooled Group (since minimal differences were expected in adverse events between participants who received different lots of the vaccine) and Flu+Placebo group. Participants that received the Flu vaccine only as standard of care (group RSV pooled) were not included for safety analyses after receiving the Flu vaccine, as this was not a study objective.
Arm/Group | RSV lot1 Group | RSV lot2 Group | RSV lot3 Group | RSV+Flu Pooled Group | Flu+Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/220 | 0/223 | 0/218 | 0/438 | 0/440
Serious Adverse Events (participants affected / at risk) | 2/220 | 1/223 | 2/218 | 4/438 | 4/440
Other Adverse Events (participants affected / at risk) | 182/220 | 193/223 | 194/218 | 409/438 | 396/440
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RSV lot1 Group (N=220) | RSV lot2 Group (N=223) | RSV lot3 Group (N=218) | RSV+Flu Pooled Group (N=438) | Flu+Placebo Group (N=440)
Joint ankylosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Greater trochanteric pain syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Multiple fractures (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cervical dysplasia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Optic neuropathy (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RSV lot1 Group (N=220) | RSV lot2 Group (N=223) | RSV lot3 Group (N=218) | RSV+Flu Pooled Group (N=438) | Flu+Placebo Group (N=440)
Administration site pain (General disorders) | 108 (108) | 131 (131) | 115 (115) | 360 (440) | 327 (346)
Fatigue (General disorders) | 110 (112) | 113 (113) | 121 (123) | 263 (268) | 230 (233)
Administration site swelling (General disorders) | 9 (9) | 11 (11) | 10 (10) | 32 (35) | 14 (14)
Administration site erythema (General disorders) | 10 (10) | 9 (9) | 10 (10) | 18 (19) | 7 (7)
Pyrexia (General disorders) | 6 (6) | 3 (3) | 8 (8) | 14 (14) | 3 (3)
Axillary pain (General disorders) | 4 (4) | 5 (5) | 4 (4) | 6 (6) | 2 (3)
Swelling (General disorders) | 5 (5) | 1 (1) | 1 (1) | 3 (3) | 1 (1)
Injection site pain (General disorders) | 4 (4) | 1 (1) | 0 (0) | 1 (1) | 5 (5)
Injection site lymphadenopathy (General disorders) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 2 (3)
Discomfort (General disorders) | 1 (1) | 0 (0) | 2 (4) | 4 (5) | 3 (3)
Pain (General disorders) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Chills (General disorders) | 0 (0) | 2 (2) | 0 (0) | 6 (6) | 1 (1)
Malaise (General disorders) | 0 (0) | 2 (2) | 0 (0) | 3 (4) | 1 (1)
Injection site pruritus (General disorders) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Injection site haematoma (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Injection site swelling (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Administration site warmth (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Injection site discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site extravasation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vaccination site haematoma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vaccination site rash (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Feeling hot (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site erythema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Temperature regulation disorder (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vaccination site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 110 (122) | 108 (115) | 108 (111) | 227 (247) | 196 (209)
Migraine (Nervous system disorders) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 3 (3)
Dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Idiopathic intracranial hypertension (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness exertional (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 34 (35) | 31 (32) | 32 (33) | 68 (72) | 54 (56)
Diarrhoea (Gastrointestinal disorders) | 29 (29) | 25 (27) | 28 (28) | 59 (64) | 77 (77)
Abdominal pain (Gastrointestinal disorders) | 25 (25) | 33 (33) | 25 (25) | 61 (61) | 63 (64)
Vomiting (Gastrointestinal disorders) | 7 (7) | 5 (5) | 3 (3) | 9 (9) | 11 (11)
Flatulence (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Frequent bowel movements (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Haemorrhoids thrombosed (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia oral (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Volvulus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 4 (4) | 4 (4) | 2 (2) | 13 (13) | 15 (15)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 0 (0) | 3 (3) | 8 (8) | 2 (3)
COVID-19 (Infections and infestations) | 0 (0) | 2 (2) | 4 (4) | 7 (7) | 2 (2)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 3 (3)
Sinusitis (Infections and infestations) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 2 (2)
Influenza (Infections and infestations) | 3 (3) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 3 (3)
Pharyngotonsillitis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Tonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Nasal herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eczema impetiginous (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Bacterial vulvovaginitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fungal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Otitis media acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Respiratory tract infection bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Suspected COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bacterial vaginosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Otitis externa (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Streptococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3) | 5 (5) | 6 (6) | 6 (6)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 1 (1) | 8 (8) | 6 (6)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 4 (4) | 3 (3) | 5 (5)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (4) | 2 (2) | 6 (6) | 4 (4)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
Catarrh (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary calcification (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4) | 1 (1) | 4 (4) | 5 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 1 (1) | 3 (3) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 4 (4) | 2 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Muscle contracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Torticollis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Axillary mass (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 6 (6) | 7 (8) | 5 (5) | 6 (6) | 4 (4)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 1 (1)
External ear inflammation (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Excessive cerumen production (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eustachian tube disorder (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Limb injury (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lip injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Patella fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thermal burn (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Animal bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fascial rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle strain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Menstrual disorder (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Heavy menstrual bleeding (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intermenstrual bleeding (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Menstruation irregular (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Menopausal symptoms (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4)
Eye symptom (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eczema eyelids (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blepharitis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bladder pain (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Body temperature increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood pressure decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Smear cervix abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
High risk sexual behaviour (Social circumstances) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Food allergy (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Immunisation reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Supernumerary teeth (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-05-26): https://cdn.clinicaltrials.gov/large-docs/44/NCT05045144/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-09): https://cdn.clinicaltrials.gov/large-docs/44/NCT05045144/SAP_001.pdf